CLINICAL TRIAL: NCT00551889
Title: Phase I Trial of Oral Cyclophosphamide in Combination With Celecoxib in Patients With Advanced Malignancies
Brief Title: Cyclophosphamide and Celecoxib in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 00191; P30CA033572 (NIH); CHNMC-00191; CDR0000570416 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Celecoxib; Cyclophosphamide

INTERVENTIONS:
Drug: celecoxib
Drug: cyclophosphamide
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Celecoxib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving cyclophosphamide together with celecoxib may help kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of celecoxib when given together with cyclophosphamide in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To describe the toxicities of oral cyclophosphamide when administered with escalating doses of celecoxib in patients with advanced malignancies.
* To evaluate the effects of this regimen on plasma levels of vascular endothelial growth factor.

OUTLINE: This is a dose-escalation study of celecoxib.

In the first course, patients receive oral cyclophosphamide once daily on days 1-35 and oral celecoxib twice daily on days 8-35. In all subsequent courses, patients receive oral cyclophosphamide once daily and oral celecoxib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline, periodically during treatment, and at time of tumor progression. Samples are analyzed for vascular endothelial growth factor levels and stored for future analysis of circulating DNA of angiogenic biomarkers.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven diagnosis of a malignant disease for which no satisfactory treatment exists at the time of enrollment
* Patients with brain metastases that, at the time of study enrollment, are controlled and do not require treatment with corticosteroids are eligible

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 3 months
* ANC > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Creatinine clearance > 50 mL/min
* Serum bilirubin < 1.5 mg/dL
* AST or ALT < 2.0 times upper limit of normal (unless clearly due to the presence of tumor)
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Patient must be capable of understanding the nature of the trial and must give written informed consent
* No unstable or severe intercurrent medical conditions or active, uncontrolled infection
* No history of allergic reactions to nonsteroidal anti-inflammatory drugs
* No bleeding peptic ulcer within the past 3 months
* No allergy to sulfa drugs

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* No radiotherapy or chemotherapy within the 3 weeks (nitrosoureas or mitomycin C within 6 weeks) prior to anticipated first day of dosing
* No concurrent therapy with other investigational agents or antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2001-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Toxicity
Maximum tolerated dose
Survival
Time to failure

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw W. Twardowski, MD, Study Chair — City of Hope Comprehensive Cancer Center